CLINICAL TRIAL: NCT02507427
Title: Safety and Efficacy of Pelvic Autonomic Nerve Monitoring and Mapping During Robot Assisted Laparoscopic Radical Prostatectomy for Preservation of Erectile Function
Brief Title: Monitoring and Mapping of Erectile Nerve During RALP (MMEN Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chang Wook Jeong, Seoul National University Hospital, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1504-070-664
Record Dates: First submitted 2015-07-22; First posted 2015-07-24 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer, robot, nerve mapping and monitoring
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nerve monitoring arm (Experimental): They will receive pelvic autonomic nerve monitoring and mapping using NIM-Eclipse (Medtronic) during robot-assisted laparoscopic prostatectomy.
  Interventions: Device: NIM-Eclipse

INTERVENTIONS:
Device: NIM-Eclipse — Using NIM-Eclipse, nerve monitoring and mapping are performed

SUMMARY:
To evaluate the safety and efficacy of pelvic autonomic nerve monitoring and mapping during robot assisted laparoscopic radical prostatectomy for preservation of erectile function.

DETAILED DESCRIPTION:
Using NIM-Eclipse monitoring instrument (Medtronic), we will check action potential of cavernous nerve, bulbocavernosus reflex and pudendal nerve somatosensory evoked potential in real time during robot assisted laparoscopic radical prostatectomy for preservation of erectile function. In this feasibility and protocol setting phase I/II study, we will evaluate the safety and efficacy of pelvic autonomic nerve monitoring and mapping using NIM-Eclipse monitoring instrument.

ELIGIBILITY:
Inclusion Criteria:

* pathologically proven localized prostate cancer (≤cT3a)
* patients to undergo robot-assisted laparoscopic prostatectomy at our center

Exclusion Criteria:

* prior hormone therapy
* prior radiation treatment on prostate or pelvis
* refused to participate

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-26 (Actual); Primary Completion 2017-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Completion rate of nerve monitoring and mapping during RALP | During the operation
  Completion rate of planed surgery without significant intra-operative complication

SECONDARY OUTCOMES:
Adverse event | 12 months
  Rate of adverse events during and after procedures upto 12 months
Quantification of erectile nerve preservation | During the operation
  Changes in action potential after prostate removal from the baseline. Electrical stimulation will be given at each neurovascular bundle 3 times. Action potential will be measured at both corpus cavernosum.
Correlation between the quantification and subjective nerve preservation grade | During the operation
  Mean value of the quantification by nerve preservation grade (Tewari et al, 2011) which was subjectively scored by the surgeon.
Correlation between the quantification of erectile nerve preservation and the postoperative recovery of erectile function | 12 months
  Recovery duration of erection measured by the International Index of Erectile Dysfunction(IIEF)-5 score according to the quantification of erectile nerve preservation

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, M.D., Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
No part of IPD will be shared.